CLINICAL TRIAL: NCT00865046
Title: Efficacy of Periosteal Stimulation and Boosters for Advanced Knee OA Pain
Brief Title: Periosteal Stimulation for Knee Osteoarthritis
Acronym: PST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A6614-R
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Osteoarthritis, Knee
Keywords: acupuncture
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PST + PST boosters (Experimental): PST once a week for 10 weeks, then tapering over 6 months
  Interventions: Other: Periosteal stimulation
- PST + control-PST boosters (Active Comparator): PST once a week for 10 weeks, then control-PST tapering over 6 months
  Interventions: Other: Periosteal stimulation; Other: Control-Periosteal Stimulation
- Control-PST (Placebo Comparator): control-PST for 10 weeks
  Interventions: Other: Control-Periosteal Stimulation

INTERVENTIONS:
Other: Periosteal stimulation — Four acupuncture needles are placed around the knee to the level of the periosteum and two needles are placed pretibially in the soft tissue. All needles are stimulated with 100 Hz current. The stimulation of the needles in the soft tissue is discontinued after one minute.
  Arms: PST + PST boosters; PST + control-PST boosters
Other: Control-Periosteal Stimulation — Acupuncture needles are placed as per the PST intervention, but only the soft tissue needles receive electrical stimulation for one minute.
  Arms: Control-PST; PST + control-PST boosters

SUMMARY:
185 veterans with chronic knee pain and advanced knee osteoarthritis will be recruited to participate in this study designed to test the effectiveness of a special type of electrical acupuncture called periosteal stimulation (PST). Participants will be divided into three groups. They will receive PST or a control condition once a week for 10 weeks. Two-thirds of the participants will receive booster sessions periodically over the course of the next 6 months. Everyone will be called monthly during the 6 month period and then will be asked to return for an evaluation on site at the end of this period.

DETAILED DESCRIPTION:
We have performed a promising initial trial of periosteal stimulation (PST, that is, electrical stimulation of 4 acupuncture needles around the knee that touch periosteum) as an analgesic for older veterans with advanced knee osteoarthritis (OA) and daily pain. The primary aim of the proposed trial is to optimize and sustain the efficacy of PST for reducing pain in veterans with advanced knee OA and unrelieved pain by combining it with booster PST. Our secondary aims are to 1) improve physical performance in these individuals, and 2) ascertain the physical and psychological predictors of response to PST. In a randomized controlled clinical trial, 180 veterans (age 50 and older) with persistent knee pain who have x-ray evidence of advanced OA will be assigned to one of three intervention groups: 1) control PST once a week for 10 weeks (i.e., needle placement with brief stimulation of non-periosteal needles), 2) PST once a week for 10 weeks followed by tapering PST boosters over 6 months, or 3) PST once a week for 10 weeks followed by tapering control-PST boosters over 6 months. Prior to initiating the intervention, immediately after the last session, and 6 months later, the following parameters will be assessed: 1) pain severity (WOMAC), 3) physical performance (gait velocity, stair climb, repetitive chair rise, timed up and go), and 4) psychological function (mood, coping, self-efficacy). Monthly telephone calls will assess pain, interim illness and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* English speaking,
* Knee pain on most days of the past 3 months that is more severe than pain in other parts of the lower body,
* Advanced knee OA by x-ray,
* age 50-89

Exclusion Criteria:

* Non-ambulatory or severely impaired mobility (i.e., require the use of a walker),
* Folstein MMSE < 24,
* Severe uncorrected visual or hearing impairment,
* Knee pain due to factors other than OA,
* Large knee effusion,
* History of corticosteroid or hyaluronic acid injection in the affected knee(s) during the preceding 3 months,
* Acute or terminal illness,
* Immune suppression,
* Anticoagulation therapy,
* Pacemaker,
* Prior PST treatment
* Active participation in other studies currently
* Age >89

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2009-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra K. Weiner, MD, Principal Investigator — Geriatric Research, Education, and Clinical Center
Locations (1):
- Geriatric Research, Education, and Clinical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Weiner DK, Moore CG, Morone NE, Lee ES, Kent Kwoh C. Efficacy of periosteal stimulation for chronic pain associated with advanced knee osteoarthritis: a randomized, controlled clinical trial. Clin Ther. 2013 Nov;35(11):1703-20.e5. doi: 10.1016/j.clinthera.2013.09.025. Epub 2013 Nov 1. PMID 24184053

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: PST once a week for 10 weeks, then tapering over 6 months
  Periosteal stimulation: Four acupuncture needles are placed around the knee to the level of the periosteum and two needles are placed pretibially in the soft tissue. All needles are stimulated with 100 Hz current. The stimulation of the needles in the soft tissue is discontinued after one minute.
- Arm 2: PST once a week for 10 weeks, then control-PST tapering over 6 months
  Periosteal stimulation: Four acupuncture needles are placed around the knee to the level of the periosteum and two needles are placed pretibially in the soft tissue. All needles are stimulated with 100 Hz current. The stimulation of the needles in the soft tissue is discontinued after one minute.
  Control-Periosteal Stimulation: Acupuncture needles are placed as per the PST intervention, but only the soft tissue needles receive electrical stimulation for one minute.
- Arm 3: control-PST for 10 weeks
  Control-Periosteal Stimulation: Acupuncture needles are placed as per the PST intervention, but only the soft tissue needles receive electrical stimulation for one minute.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3
Started | 63 | 64 | 63
Completed | 57 | 59 | 62
Not Completed | 6 | 5 | 1
Not completed — Lost to Follow-up | 1 | 4 | 0
Not completed — Death | 0 | 1 | 1
Not completed — Withdrawal by Subject | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Community dwelling adults with advanced knee osteoarthritis and chronic pain
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Total
Number analyzed (Participants) | 63 | 64 | 63 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (8.9) | 65.8 (8.7) | 66.8 (10.4) | 66.5 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 11 | 29
  Male | 55 | 54 | 52 | 161
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 61 | 64 | 63 | 188
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 18 | 22 | 16 | 56
  White | 45 | 42 | 47 | 134
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 63 | 64 | 63 | 190
WOMAC [Mean (Standard Deviation); unit: units on a scale] — The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) consists of 24 items divided into 3 subscales:
  Pain (5 items), score range 0-20 Stiffness (2 items): score range 0-8 Physical Function (17 items): score range 0-68 Total score ranges from 0 (best possible outcome) to 96 (worst possible outcome)
  units on a scale | 9.0 (3.2) | 9.9 (4.0) | 10.6 (3.6) | 9.8 (3.6)
Short Physical Performance Battery [Mean (Standard Deviation); unit: units on a scale] — The SPPB measures performance on 3 items:
  1. Repeated chair stands (number of stands and time to complete as well as a 0-4 ordinal scale))
  2. Balance testing - semitandem stand, side-by-side stand, and tandem stand; each scored as 2 (held for 10 sec), 1 (held for less than 10 sec), 0 (not attempted) as well as a 0-4 ordinal scale for overall balance performance
  3. 8 foot walk - 0-4 scale according to velocity Summary ordinal score: 0 (worst performance) to 12 (best performance)
  units on a scale | 6.1 (1.8) | 6.1 (1.9) | 6.2 (1.5) | 6.1 (1.7)
Timed stair climb [Mean (Standard Deviation); unit: seconds] — Participants were timed as they ascended and descended 5 steps.
  seconds | 12.5 (4.7) | 14.5 (7.8) | 13.9 (7.3) | 13.6 (6.6)
Timed Up and Go [Mean (Standard Deviation); unit: seconds] — The Timed Up and Go (TUG) measures mobility and falls risk. The participant sits in a chair and is timed as (s)he stands up from the chair, walks 3 meters, turns around, walks back to the chair and sits down. The result is expressed in seconds. An older adult who takes at least 12 seconds to complete the TUG is at high risk for falling.
  seconds | 12.3 (3.4) | 13.1 (3.8) | 13.9 (6.9) | 13.1 (4.7)
CES-D [Mean (Standard Deviation); unit: units on a scale] — The Center for Epidemiological Studies-Depression (CES-D) scale is a measure of depressive symptoms. It is a 20 item. Each item is scored from 0 (rarely or none of the time) to 3 (most or all of the time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
  units on a scale | 11.7 (10.3) | 14.7 (11.2) | 12.3 (9.6) | 12.9 (10.4)
Cognitive Strategies Questionnaire, catastrophizing scale [Mean (Standard Deviation); unit: units on a scale] — The catastrophizing scale of the Cognitive Strategies Questionnaire consists of 6 items, each scored from 0 (never state that) to 6 (always state that). The scoring range on the instrument is 0 (best pain coping) to 36 (worst pain coping).
  units on a scale | 7.9 (7.8) | 12.1 (9.7) | 8.8 (9.2) | 9.6 (8.9)
BMI [Mean (Standard Deviation); unit: kg/m2] | 31.6 (6.5) | 33.1 (6.2) | 32.5 (6.9) | 32.4 (6.5)
Mean number of pain medications [Mean (Standard Deviation); unit: medication] — Mean number of pain medications per day
  medication | 1.1 (1.0) | 1.2 (0.9) | 1.0 (0.9) | 1.1 (0.9)
Mean number of opioids [Mean (Standard Deviation); unit: opioids] — Mean number of opioids per day
  opioids | 0.1 (0.3) | 0.3 (0.6) | 0.2 (0.4) | 0.2 (0.4)
Duration of knee pain [Mean (Standard Deviation); unit: years] | 5.7 (6.4) | 6.2 (6.8) | 7.2 (8.3) | 6.4 (7.2)
Arthritis Self-Efficacy score, pain [Mean (Standard Deviation); unit: units on a scale] — This is the pain subscale of The Arthritis Self-Efficacy Scale (ASES). The ASES consists of 20 questions divided into three subscales: physical function (9 questions), other symptoms (6 questions) and pain (5 questions). Participants are asked about their level of certainty that they can perform each task. Each question is scored from 10 = very uncertain to 100 = very certain. Each subscale is scored separately by taking the mean score of the items. Higher scores indicate higher self-efficacy. The range for the pain subscale is 10 to 100.
  units on a scale | 64.3 (21.6) | 59.5 (22.6) | 63.9 (21.7) | 62.6 (22)
Arthritis Self-Efficacy score, function [Mean (Standard Deviation); unit: units on a scale] — This is the physical function subscale of The Arthritis Self-Efficacy Scale (ASES). The ASES consists of 20 questions divided into three subscales: physical function (9 questions), other symptoms (6 questions) and pain (5 questions). Participants are asked about their level of certainty that they can perform each task. Each question is scored from 10 = very uncertain to 100 = very certain. Each subscale is scored separately by taking the mean score of the items. Higher scores indicate higher self-efficacy. The range for the physical function subscale is 10 to 100.
  units on a scale | 77.5 (17.0) | 76.3 (16.9) | 76.1 (16.4) | 76.6 (16.8)
Arthritis Self-Efficacy score, other symptoms [Mean (Standard Deviation); unit: units on a scale] — This is the other symptoms subscale of The Arthritis Self-Efficacy Scale (ASES). The ASES consists of 20 questions divided into three subscales: physical function (9 questions), other symptoms (6 questions) and pain (5 questions). Participants are asked about their level of certainty that they can perform each task. Each question is scored from 10 = very uncertain to 100 = very certain. Each subscale is scored separately by taking the mean score of the items. Higher scores indicate higher self-efficacy. The range for the other symptoms subscale is 10 to 100.
  units on a scale | 70.5 (21.1) | 65.9 (20.3) | 68.6 (20.9) | 68.3 (20.8)

OUTCOME MEASURES:

1. Primary Outcome: Pain (WOMAC)
Description: The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) consists of 24 items divided into 3 subscales:
  Pain (5 items), score range 0-20 Stiffness (2 items): score range 0-8 Physical Function (17 items): score range 0-68 Total score ranges from 0 (best possible outcome) to 96 (worst possible outcome)
Time Frame: 9 months following baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 57 | 59 | 62
units on a scale | 6.1 (3.5) | 6.6 (3.6) | 7.9 (7.7)

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2 | Arm 3
Serious Adverse Events (participants affected / at risk) | 3/63 | 1/64 | 1/63
Other Adverse Events (participants affected / at risk) | 3/63 | 0/64 | 1/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=63) | Arm 2 (N=64) | Arm 3 (N=63)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) — The participant completed participation in the trial. This participant was scheduled to undergo a one year follow-up questionnaire in 6-11 and died 3-11-11.
Bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=63) | Arm 2 (N=64) | Arm 3 (N=63)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
sweating (General disorders) | 0 (0) | 0 (0) | 0 (0)
Lightheaded (General disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes